CLINICAL TRIAL: NCT07086274
Title: Efficacy of Individualized Location-based Repetitive Transcranial Magnetic Stimulation in the Treatment of Migraine: a Prospective Clinical Study
Brief Title: Individualized Location-based rTMS for Migraine Treatment: A Multicenter Clinical Study
Acronym: individua rTMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: The Affiliated Hospital of Hangzhou Normal University (Other); Red Cross Hospital, Hangzhou, China (Other); The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: [2025C]IIT. No. 013
Record Dates: First submitted 2025-03-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-03

CONDITIONS: Migraine; Transcranial Magnetic Stimulation Repetitive
Keywords: Individualized location-based
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized location-based Repetitive Transcranial Magnetic Stimulation (Experimental): Enhancing targeting accuracy through personalized target localization to improve the analgesic response rate of rTMS.
  Interventions: Device: Individualized location-based Repetitive Transcranial Magnetic Stimulation
- Traditional location-based Repetitive Transcranial Magnetic Stimulation (Active Comparator): Recent studies have shown that the dorsolateral prefrontal cortex (DLPFC) plays an inhibitory role in the human pain pathway. High-frequency repetitive transcranial magnetic stimulation (rTMS) applied to the left DLPFC has been found to improve chronic migraine.
  Interventions: Device: Traditional location-based Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Individualized location-based Repetitive Transcranial Magnetic Stimulation — Enhancing targeting accuracy through personalized target localization to improve the analgesic response rate of rTMS.
  Arms: Individualized location-based Repetitive Transcranial Magnetic Stimulation
Device: Traditional location-based Repetitive Transcranial Magnetic Stimulation — Recent studies have shown that the dorsolateral prefrontal cortex (DLPFC) plays an inhibitory role in the human pain pathway. High-frequency repetitive transcranial magnetic stimulation (rTMS) applied to the left DLPFC has been found to improve chronic migraine.
  Arms: Traditional location-based Repetitive Transcranial Magnetic Stimulation

SUMMARY:
For migraine patients experiencing at least four attack days per month and undergoing transcranial magnetic stimulation (TMS) treatment, a randomized, double-blind controlled trial is conducted, dividing participants into a traditional targeting group and an individualized targeting group. Patients in both groups are followed up before treatment and at 1, 2, and 3 months post-treatment, evaluating the following parameters: migraine diaries, the number of migraine days, rescue medication usage, headache intensity, the number of moderate-to-severe migraine days, and the proportion of patients achieving a ≥50% reduction in migraine days. Further assessments include changes in the Migraine Disability Assessment (MIDAS), Headache Impact Test-6 (HIT-6), Migraine-Specific Quality of Life Questionnaire (MSQ), Pittsburgh Sleep Quality Index (PSQI), Patient Global Impression of Change (PGIC), 24-item Hamilton Depression Scale (HAMD-24), and 14-item Hamilton Anxiety Scale (HAMA-14). Biomarker and metabolic analyses include tryptophan and kynurenine metabolism, calcitonin gene-related peptide (CGRP), pituitary adenylate cyclase-activating polypeptide (PACAP), vasoactive intestinal peptide (VIP), neuropeptide Y (NPY), substance P, endothelin-1, inflammatory cytokines (IL-1β, IL-6, TNF-α, TGF-β1), glutamate, endocannabinoids and related lipids, as well as gut microbiota composition. Additionally, changes in resting-state functional magnetic resonance imaging (rs-fMRI) before and after treatment are analyzed. This study aims to compare the efficacy of TMS treatment under different targeting strategies in migraine patients, providing theoretical support for clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years; both men and women.
* Diagnosis of migraine according to the International Classification of Headache Disorders, 3rd edition (ICHD-III), with first onset before age 50 and a history of migraine for more than 1 year.
* Migraine frequency of ≥4 days per month during both the 3 months prior to the screening period and the screening period itself.
* Informed consent documents are signed, and subjects are cooperative with the evaluation and rTMS treatment, having been informed of known and potential risks and available alternative treatments.

Exclusion Criteria:

* Patients with contraindications to TMS (e.g., metal implants, pacemakers).
* Severe anxiety or depression (HAMD score >35, HAMA score >29).
* History of migraine prophylactic drug adjustment during the screening and treatment period.
* Aphasia or cognitive dysfunction (MMSE score ≤23).
* Pregnancy or lactation.
* Clinicians assess severe comorbidities that are not treatable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2027-07-25 (Estimated); Study Completion 2027-07-25 (Estimated)

PRIMARY OUTCOMES:
Change in the monthly average number of migraine days | from baseline to 1 month after treatment completion.
  A migraine day: any calendar day in which the participant experienced a qualified migraine headache (onset, continuation, or recurrence of the migraine headache). A qualified migraine headache: a migraine with or without aura, lasting for ≥30 minutes, and meeting at least 1 of the following criteria (a and/or b): a) ≥2 of the following: unilateral location, pulsating quality, moderate to severe pain intensity, aggravation by or causing avoidance of routine physical activity; b) ≥1 of the following: nausea and/or vomiting, photophobia, and phonophobia. If the participant took a migraine-specific medication during aura or to treat headache on a calendar day, it was counted as a migraine day regardless of the duration and pain features/associated symptoms.

SECONDARY OUTCOMES:
Change in the monthly average number of migraine days | from baseline to 2.3 month after treatment completion.
  A migraine day was any calendar day in which the participant experienced a qualified migraine headache (as previously described). If the participant took a migraine-specific medication during aura or to treat headache on a calendar day, it was counted as a migraine day regardless of the duration and pain features/associated symptoms. A moderate or severe migraine day was a migraine day of moderate or severe pain intensity. Months were defined as 28-day intervals.
Mean Change From Baseline in the Migraine Disability Assessment (MIDAS) Total Score | Compared to baseline 3 months after treatment completion.
  The Migraine Disability Assessment (MIDAS) is a retrospective, self-administered, 5-item questionnaire that measures headache-related disability as lost time due to headache from paid work or school, household work, and non-work activities. Participants provide the number of missed work or school days; missed household chores days; missed social or leisure activity days; and days at work or school, and separately at home, where productivity was reduced by half or more in the last 3 months (scale: 0 - 90 for each of 5 subscales). The 5 subscale scores are summed to compute the MIDAS total score (scale: 0 - 450). Lower scores indicate less headache-related disability.
Mean Change From Baseline in the Migraine-Specific Quality of Life Questionnaire (MSQ) | from baseline to 1.2.3 month after treatment completion.
  The Migraine Specific Quality of Life (MSQoL) is a self-administered, 14-item instrument that has been validated in 3 domains: role restriction, role prevention, and the emotional function. The role function-restrictive domain consists of 7 items that describe how migraine limits one's daily social and work-related activities. Participants respond to items using a 6-point scale: "none of the time," "a little bit of the time," "some of the time," "a good bit of the time," "most of the time," and "all of the time," which are assigned scores of 1 to 6, respectively. Item scores are recoded using (7 - original score). Next, raw dimension scores are computed as a sum of recoded item scores and rescaled from a 0 to 100 scale such that higher scores indicate better quality of life.
Mean Change From Baseline in the Headache Impact Test-6 (HIT-6 ) | from baseline to 1.2.3 month after treatment completion.
  HIT-6 (Headache Impact Test-6) for Migraine: The HIT-6 is a widely used tool to assess the impact of headaches on a patient's quality of life. It consists of 6 questions, each rated on a 5-point scale ranging from "Never" to "Always." The total score is obtained by summing the individual item scores, with a higher score indicating a greater impact of migraine on the patient's daily functioning. A decrease in the HIT-6 score from baseline indicates an improvement in the patient's condition and a reduction in the impact of migraines on their life.
Mean Change From Baseline in the Pittsburgh Sleep Quality Index(PSQI ) | from baseline to 1.2.3 month after treatment completion.
  PSQI (Pittsburgh Sleep Quality Index) for Sleep: The PSQI is a validated questionnaire used to assess the quality and patterns of sleep in the past month. It includes 19 items across 7 component areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is scored on a 0 to 3 scale, and the total score ranges from 0 to 21, with higher scores indicating poorer sleep quality. A decrease in the PSQI score from baseline indicates an improvement in sleep quality.
Mean Change From Baseline in the Patient Global Impression of Change(PGIC ) | from baseline to 3 month after treatment completion.
  PGIC (Patient Global Impression of Change): The PGIC is a single-item scale used to assess the patient's overall perception of change in their condition over time. The patient rates their perceived change in symptoms or overall health since the start of the study or treatment on a 7-point scale, where:
  1. = Very Much Improved
  2. = Much Improved
  3. = Minimally Improved
  4. = No Change
  5. = Minimally Worse
  6. = Much Worse
  7. = Very Much Worse
  A higher score indicates a negative change in the patient's condition, while a lower score indicates improvement. The mean change from baseline reflects the overall perceived improvement or worsening of the patient's condition during the study period.
Mean Change From Baseline in the HAMD-24 (Hamilton Depression Rating Scale, 24-item). | from baseline to 1.2.3 month after treatment completion.
  HAMD-24 (Hamilton Depression Rating Scale, 24-item): The HAMD-24 is a clinician-administered scale used to assess the severity of depressive symptoms. It consists of 24 items, with each item scored on a 3 to 5-point scale based on the severity of the symptom (e.g., 0 = not present, 1 = mild, 2 = moderate, 3 = severe). The total score is calculated by summing the individual item scores, with higher scores indicating more severe depression. A reduction in the HAMD-24 score from baseline indicates improvement in the severity of depressive symptoms.
Mean Change From Baseline in the HAMA-14 (Hamilton Anxiety Rating Scale, 14-item). | from baseline to 1.2.3 month after treatment completion.
  HAMA-14 (Hamilton Anxiety Rating Scale, 14-item): The HAMA-14 is a clinician-administered scale used to assess the severity of anxiety symptoms. It includes 14 items that cover both psychic and somatic aspects of anxiety, such as tension, fear, insomnia, and somatic symptoms (e.g., gastrointestinal distress, dizziness). Each item is rated on a 5-point scale ranging from 0 (not present) to 4 (severe). The total score is calculated by summing the individual item scores, with higher scores indicating greater severity of anxiety. A reduction in the HAMA-14 score from baseline indicates a decrease in anxiety symptoms.
Metabolomics (Tryptophan and Kynurenine) | Treatment completion (2 weeks) vs. baseline.
  Tryptophan and Kynurenine:
  Measurement Method: Liquid Chromatography-Mass Spectrometry (LC-MS) or High-Performance Liquid Chromatography (HPLC) with UV detection.
  Units: µmol/L or nmol/mL.
Mean Change From Baseline in Inflammatory Biomarker Levels. | Treatment completion (2 weeks) vs. baseline.
  CGRP (Calcitonin Gene-Related Peptide), PACAP (Pituitary Adenylate Cyclase-Activating Polypeptide), VIP (Vasoactive Intestinal Peptide), NPY (Neuropeptide Y), Substance P, Endothelin-1:
  Measurement Method: Enzyme-Linked Immunosorbent Assay (ELISA), Radioimmunoassay (RIA), or Luminex xMAP technology.
  Units: pg/mL or ng/mL.
  Inflammatory Factors (IL-1β, IL-6, TNF-α, TGF-β1):
  Measurement Method: ELISA. Units: pg/mL or ng/mL.
Mean Change From Baseline in Glutamate, Endocannabinoids and Related Lipids | Treatment completion (2 weeks) vs. baseline.
  Glutamate:
  Measurement Method:High-Performance Liquid Chromatography (HPLC) with fluorescence detection or LC-MS/MS.
  Units:µmol/L or nmol/mL.
  Endocannabinoids:
  Measurement Method:Liquid Chromatography-Mass Spectrometry (LC-MS) or Gas Chromatography-Mass Spectrometry (GC-MS).
  Units: pg/mL or nmol/L.
  Related Lipids:
  Measurement Method: LC-MS/MS or Gas Chromatography-Mass Spectrometry (GC-MS). Units:ng/mL or µg/mL.
Mean Change From Baseline in Gut Microbiota Composition | Treatment completion (2 weeks) vs. baseline.
  Gut Microbiota:
  Measurement Method: 16S rRNA Gene Sequencing (Next-Generation Sequencing, NGS) or Metagenomic Sequencing.
  Units: Relative abundance (percentage of total microbiota composition) or Operational Taxonomic Unit (OTU) counts.
Changes in pain-related brain regions and connectivity in resting-state functional magnetic resonance imaging (rs-fMRI) | Treatment completion (2 weeks) vs. baseline.
  Resting-State fMRI (rs-fMRI): This imaging technique assesses brain activity in the absence of an explicit task. It measures spontaneous fluctuations in the blood oxygen level-dependent (BOLD) signal, which is an indicator of neural activity.
  Analysis Focus:The primary focus is on pain-related brain regions such as the somatosensory cortex, anterior cingulate cortex (ACC), insula, thalamus, and prefrontal cortex , as well as changes in the functional connectivity between these regions.
  Connectivity Analysis:Functional connectivity will be evaluated by examining seed-based analysis or independent component analysis (ICA) to identify altered networks related to pain processing and perception.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: mar-15-2025. jun-15-2027